CLINICAL TRIAL: NCT01243372
Title: Evaluating BRAF Mutations as Predictors of Efficacy in Cetuximab-Treated Colorectal Cancer Patients: A Retrospective Study of Tissues From CALGB / SWOG
Brief Title: Biomarkers in Predicting Response to Cetuximab in Patients With Advanced Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-SWOG-150506-80405-BRAF; CALGB-SWOG-150506-80405-BRAF; CDR0000688745 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2010-11-17; First posted 2010-11-18 (Estimated); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Colorectal Cancer
Keywords: recurrent colon cancer; stage IIIA colon cancer; stage IIIB colon cancer; stage IIIC colon cancer; stage IVA colon cancer; stage IVB colon cancer; recurrent rectal cancer; stage III rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Correlative (BRAF V600E mutation analysis): Previously collected formalin-fixed and paraffin-embedded baseline tumor samples are analyzed for BRAF V600E mutation. Mutation status is correlated with clinical response and outcome data from patients enrolled on CALGB-C80405.
  Interventions: Genetic: mutation analysis; Other: laboratory biomarker analysis

INTERVENTIONS:
Genetic: mutation analysis
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tissue in the laboratory from patients who received cetuximab may help doctors understand and predict how well patients will respond to treatment.

PURPOSE: This research study is studying biomarkers in predicting response to cetuximab in patients with advanced colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine, among patients with advanced CRC, whether the effect of treatment (cetuximab vs bevacizumab) on progression-free survival (PFS) depends on tumor BRAF V600E mutational status.

Secondary

* To study the relationships between tumor BRAF V600E mutational status, OS, and tumor response.

OUTLINE: This is a multicenter study.

Previously collected formalin-fixed and paraffin-embedded baseline tumor samples are analyzed for BRAF V600E mutation. Mutation status is correlated with clinical response and outcome data from patients enrolled on CALGB-C80405.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Participation in CALGB-C80405

  * Have KRAS WT or KRAS mut tumor
  * Randomized to treatment with either bevacizumab or cetuximab alone

    * Patients randomized to the combination therapy are not eligible
* Available specimens at the PCO for BRAF mutation detection
* Patient consent for use of samples

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients previously enrolled on CALGB-C80405 who have KRAS WT or KRAS mut tumor and have been randomized to treatment with either bevacizumab or cetuximab alone in a primary care clinic setting.
Sampling Method: Probability Sample
Enrollment: 1142 (Estimated)
Dates: Start 2009-11 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Progression-free survival as measured by RECIST | Up to 36 months

SECONDARY OUTCOMES:
overall survival | Up to 36 months
tumor response as measured by RECIST | Up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Najjia N. Mahmoud, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine